CLINICAL TRIAL: NCT04675073
Title: Preventive VT Substrate Ablation in Patients With Chronic Post-MI Scar Showing Arrhythmogenic Characteristics
Brief Title: Preventive VT Substrate Ablation in Ischemic Heart Disease
Acronym: PREVENT-VT
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centro Medico Teknon (Other)
Responsible Party: Principal Investigator, Antonio Berruezo, MD, PhD, Head of Arrhythmia Section, Centro Medico Teknon
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PREVENT-VT
Record Dates: First submitted 2020-11-29; First posted 2020-12-19 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Ventricular Tachycardia; Ventricular Arrythmia; Sudden Cardiac Death; Sudden Cardiac Death Due to Cardiac Arrhythmia; Ischemic Heart Disease; Myocardial Infarction; Magnetic Resonance Imaging
Keywords: ventricular tachycardia; ventricular arrhythmia; sudden cardiac death; ischemic heart disease; cardiac magnetic resonance; border zone channels
MeSH Terms: conditions — Tachycardia, Ventricular; Death, Sudden, Cardiac; Myocardial Ischemia; Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ABLATE arm (Experimental): Ventricular tachycardia substrate ablation intending to: i) eliminate all the potential arrhythmogenic substrate, aiming for complete electrical isolation/elimination of all the electrograms with delayed components or showing hidden slow conduction properties, and ii) non-inducibility or ventricular tachycardias at the end of the procedure. Standard medical treatment will also be given for these patients.
  Interventions: Procedure: Ventricular tachycardia substrate-based radiofrequency ablation
- NO-TREAT arm (No Intervention): Only standard medical treatment will be offered for these patients.

INTERVENTIONS:
Procedure: Ventricular tachycardia substrate-based radiofrequency ablation — The CARTO3 electroanatomic navigation system (Biosense Webster, Diamond Bar, CA, USA) will be used for ablation. An open irrigated 3.5-mm tip ablation catheter (ThermoCool SmartTouch, Biosense Webster, Diamond Bar, CA, USA) will be used for mapping and ablation. The first step of the procedure will be the acquisition of a fast-anatomical map (FAM) of the aorta. This FAM will be then used to integrate the multi-detector cardiac tomography (MDCT) reconstruction and cardiac magnetic resonance (CMR)-derived pixel-signal intensity (PSI) maps within the spatial reference coordinates of the CARTO3 system. RF will be delivered at the entrance of the border zone channels (BZCs) identified in the PSI maps (CMR-guided scar dechanneling technique). Programmed ventricular stimulation (PVS) will be always performed after substrate elimination to test for final inducibility.
  Arms: ABLATE arm

SUMMARY:
The investigators hypothesize that preventive VT substrate ablation in patients with chronic ICM, previously selected based on imaging criteria (BZC mass) for their likely high arrhythmic risk, is safe and effective in preventing clinical VT events.

DETAILED DESCRIPTION:
Fibrotic tissue is known to be the substrate for the appearance of scar-related reentrant ventricular arrhythmias (VA) in chronic ischemic cardiomyopathy (ICM). Late gadolinium enhancement cardiac magnetic resonance (LGE-CMR) has proven to be a useful technique in the non-invasive characterization of the scarred tissue and the underlying arrhythmogenic substrate. Previous studies identified the presence of significant scarring (>5% of the LV mass) is an independent predictor of adverse outcome (all-cause mortality or appropriate ICD discharge for ventricular tachycardia or fibrillation) in patients being considered for implantable cardioverter-defibrillator (ICD) placement. Parallelly, the presence of heterogeneous tissue channels, which correlate with voltage channels after endocardial voltage mapping of the scar, can be more frequently observed in patients suffering from SMVT than in matched controls for age, sex, infarct location, and LVEF. However, the lack of solid evidence and randomized trials make LVEF still the main decision parameter when assessing suitability for ICD implantation in primary prevention of SCD. (7,8) In a recent, case-control study, the investigators identified the BZC mass as the only independent predictor for VT occurrence, after matching for age, sex, LVEF and total scar mass. This BZC mass can be automatically calculated using a commercially available, post-processing imaging platform named ADAS 3D LV (ADAS3D Medical SL, Barcelona, Spain), with FDA 510(k) Clearance and CE Mark approval. Thus, CMR-derived BZC mass might be used as an automatically reproducible criterium to reclassify those patients with chronic ICM at highest risk for developing VA/SCD in a relatively short period of time (approx. 2 years).

On the other hand, catheter ablation has become an essential tool in the treatment of ventricular arrhythmias in patients with structural heart disease (SHD). VT ablation techniques have evolved towards substrate-based approaches that permit to abolish multiple VT circuits irrespective of their inducibility or hemodynamic tolerability, improving outcomes with respect to clinical VT ablation. Moreover, VT substrate ablation procedures performed during sinus rhythm and CMR-guided have proven to be safe, with very low procedure related complications.

The investigators hypothesize that preventive VT substrate ablation in patients with chronic ICM, previously selected based on imaging criteria (BZC mass) for their likely high arrhythmic risk, is safe and effective in preventing clinical VT events.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years.
* Chronic, stable ischemic heart disease, irrespectively of the LVEF.
* Life expectancy of > 1 year with a good functional status.
* Documented scar AND a BZC mass > 5.15 g as measured per LGE-CMR and automatic post-processing using the ADAS-3D LV (ADAS 3D Medical SL, Barcelona, Spain).
* Signed informed consent.

Exclusion Criteria:

* Age < 18 years.
* Pregnancy.
* Life expectancy of < 1 year, or bad functional status (NYHA IV functional class).
* Other concomitant structural heart diseases (e.g. congenital, non-ischemic, etc.)
* Previously documented sustained ventricular arrhythmias.
* Impossibility to perform a contrast-enhanced CMR study.
* Calculated BZC mass in the scarred tissue < 5.15 g using the ADAS-3D LV software.
* Concomitant investigation treatments.
* Medical, geographical and social factors that make study participation impractical, and inability to give written informed consent. Patient's refusal to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Rate of sudden cardiac death or sustained ventricular tachycardia | 2 years
  Composite outcome of sudden cardiac death or sustained ventricular tachycardia (either treated by an ICD or documented with continuous Holter monitoring) in patients undergoing preventive ventricular tachycardia (VT) substrate ablation vs. standard of care.

SECONDARY OUTCOMES:
Procedure time | 2 years
  Procedure time
Radiofrequency time | 2 years
  Radiofrequency time
Rate of achievement of complete substrate ablation | 2 years
  Rate of achievement of complete substrate ablation
VT inducibility rate | 2 years
  Final VT inducibility rate
Rate of complications | 2 years
  Rate of complications
Rate of need for anti-arrhythmic drugs | 2 years
  Rate of need for anti-arrhythmic drugs in both arms of the study

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Berruezo, MD, PhD, Principal Investigator — Centro Médico Teknon
Locations (1):
- Centro Medico Teknon, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] de Bakker JM, van Capelle FJ, Janse MJ, Wilde AA, Coronel R, Becker AE, Dingemans KP, van Hemel NM, Hauer RN. Reentry as a cause of ventricular tachycardia in patients with chronic ischemic heart disease: electrophysiologic and anatomic correlation. Circulation. 1988 Mar;77(3):589-606. doi: 10.1161/01.cir.77.3.589. PMID 3342490
- [Background] Wu E, Judd RM, Vargas JD, Klocke FJ, Bonow RO, Kim RJ. Visualisation of presence, location, and transmural extent of healed Q-wave and non-Q-wave myocardial infarction. Lancet. 2001 Jan 6;357(9249):21-8. doi: 10.1016/S0140-6736(00)03567-4. PMID 11197356
- [Background] Schmidt A, Azevedo CF, Cheng A, Gupta SN, Bluemke DA, Foo TK, Gerstenblith G, Weiss RG, Marban E, Tomaselli GF, Lima JA, Wu KC. Infarct tissue heterogeneity by magnetic resonance imaging identifies enhanced cardiac arrhythmia susceptibility in patients with left ventricular dysfunction. Circulation. 2007 Apr 17;115(15):2006-14. doi: 10.1161/CIRCULATIONAHA.106.653568. Epub 2007 Mar 26. PMID 17389270
- [Background] Yan AT, Shayne AJ, Brown KA, Gupta SN, Chan CW, Luu TM, Di Carli MF, Reynolds HG, Stevenson WG, Kwong RY. Characterization of the peri-infarct zone by contrast-enhanced cardiac magnetic resonance imaging is a powerful predictor of post-myocardial infarction mortality. Circulation. 2006 Jul 4;114(1):32-9. doi: 10.1161/CIRCULATIONAHA.106.613414. Epub 2006 Jun 26. PMID 16801462
- [Background] Klem I, Weinsaft JW, Bahnson TD, Hegland D, Kim HW, Hayes B, Parker MA, Judd RM, Kim RJ. Assessment of myocardial scarring improves risk stratification in patients evaluated for cardiac defibrillator implantation. J Am Coll Cardiol. 2012 Jul 31;60(5):408-20. doi: 10.1016/j.jacc.2012.02.070. PMID 22835669
- [Background] Perez-David E, Arenal A, Rubio-Guivernau JL, del Castillo R, Atea L, Arbelo E, Caballero E, Celorrio V, Datino T, Gonzalez-Torrecilla E, Atienza F, Ledesma-Carbayo MJ, Bermejo J, Medina A, Fernandez-Aviles F. Noninvasive identification of ventricular tachycardia-related conducting channels using contrast-enhanced magnetic resonance imaging in patients with chronic myocardial infarction: comparison of signal intensity scar mapping and endocardial voltage mapping. J Am Coll Cardiol. 2011 Jan 11;57(2):184-94. doi: 10.1016/j.jacc.2010.07.043. PMID 21211689
- [Background] Moss AJ, Zareba W, Hall WJ, Klein H, Wilber DJ, Cannom DS, Daubert JP, Higgins SL, Brown MW, Andrews ML; Multicenter Automatic Defibrillator Implantation Trial II Investigators. Prophylactic implantation of a defibrillator in patients with myocardial infarction and reduced ejection fraction. N Engl J Med. 2002 Mar 21;346(12):877-83. doi: 10.1056/NEJMoa013474. Epub 2002 Mar 19. PMID 11907286
- [Background] Bardy GH, Lee KL, Mark DB, Poole JE, Packer DL, Boineau R, Domanski M, Troutman C, Anderson J, Johnson G, McNulty SE, Clapp-Channing N, Davidson-Ray LD, Fraulo ES, Fishbein DP, Luceri RM, Ip JH; Sudden Cardiac Death in Heart Failure Trial (SCD-HeFT) Investigators. Amiodarone or an implantable cardioverter-defibrillator for congestive heart failure. N Engl J Med. 2005 Jan 20;352(3):225-37. doi: 10.1056/NEJMoa043399. PMID 15659722
- [Background] Sapp JL, Wells GA, Parkash R, Stevenson WG, Blier L, Sarrazin JF, Thibault B, Rivard L, Gula L, Leong-Sit P, Essebag V, Nery PB, Tung SK, Raymond JM, Sterns LD, Veenhuyzen GD, Healey JS, Redfearn D, Roux JF, Tang AS. Ventricular Tachycardia Ablation versus Escalation of Antiarrhythmic Drugs. N Engl J Med. 2016 Jul 14;375(2):111-21. doi: 10.1056/NEJMoa1513614. Epub 2016 May 5. PMID 27149033
- [Background] Di Biase L, Burkhardt JD, Lakkireddy D, Carbucicchio C, Mohanty S, Mohanty P, Trivedi C, Santangeli P, Bai R, Forleo G, Horton R, Bailey S, Sanchez J, Al-Ahmad A, Hranitzky P, Gallinghouse GJ, Pelargonio G, Hongo RH, Beheiry S, Hao SC, Reddy M, Rossillo A, Themistoclakis S, Dello Russo A, Casella M, Tondo C, Natale A. Ablation of Stable VTs Versus Substrate Ablation in Ischemic Cardiomyopathy: The VISTA Randomized Multicenter Trial. J Am Coll Cardiol. 2015 Dec 29;66(25):2872-2882. doi: 10.1016/j.jacc.2015.10.026. PMID 26718674
- [Background] Soto-Iglesias D, Penela D, Jauregui B, Acosta J, Fernandez-Armenta J, Linhart M, Zucchelli G, Syrovnev V, Zaraket F, Teres C, Perea RJ, Prat-Gonzalez S, Doltra A, Ortiz-Perez JT, Bosch X, Camara O, Berruezo A. Cardiac Magnetic Resonance-Guided Ventricular Tachycardia Substrate Ablation. JACC Clin Electrophysiol. 2020 Apr;6(4):436-447. doi: 10.1016/j.jacep.2019.11.004. Epub 2020 Feb 26. PMID 32327078
- [Background] Fernandez-Armenta J, Soto-Iglesias D, Silva E, Penela D, Jauregui B, Linhart M, Bisbal F, Acosta J, Fernandez M, Borras R, Villuendas R, Cano L, Guasch E, Mont L, Berruezo A. Safety and Outcomes of Ventricular Tachycardia Substrate Ablation During Sinus Rhythm: A Prospective Multicenter Registry. JACC Clin Electrophysiol. 2020 Oct 26;6(11):1435-1448. doi: 10.1016/j.jacep.2020.07.028. PMID 33121673
- [Background] Knuuti J, Wijns W, Saraste A, Capodanno D, Barbato E, Funck-Brentano C, Prescott E, Storey RF, Deaton C, Cuisset T, Agewall S, Dickstein K, Edvardsen T, Escaned J, Gersh BJ, Svitil P, Gilard M, Hasdai D, Hatala R, Mahfoud F, Masip J, Muneretto C, Valgimigli M, Achenbach S, Bax JJ; ESC Scientific Document Group. 2019 ESC Guidelines for the diagnosis and management of chronic coronary syndromes. Eur Heart J. 2020 Jan 14;41(3):407-477. doi: 10.1093/eurheartj/ehz425. No abstract available. PMID 31504439
- [Background] Andreu D, Ortiz-Perez JT, Fernandez-Armenta J, Guiu E, Acosta J, Prat-Gonzalez S, De Caralt TM, Perea RJ, Garrido C, Mont L, Brugada J, Berruezo A. 3D delayed-enhanced magnetic resonance sequences improve conducting channel delineation prior to ventricular tachycardia ablation. Europace. 2015 Jun;17(6):938-45. doi: 10.1093/europace/euu310. Epub 2015 Jan 23. PMID 25616406
- [Background] Andreu D, Berruezo A, Ortiz-Perez JT, Silva E, Mont L, Borras R, de Caralt TM, Perea RJ, Fernandez-Armenta J, Zeljko H, Brugada J. Integration of 3D electroanatomic maps and magnetic resonance scar characterization into the navigation system to guide ventricular tachycardia ablation. Circ Arrhythm Electrophysiol. 2011 Oct;4(5):674-83. doi: 10.1161/CIRCEP.111.961946. Epub 2011 Aug 31. PMID 21880674
- [Background] Acosta J, Fernandez-Armenta J, Penela D, Andreu D, Borras R, Vassanelli F, Korshunov V, Perea RJ, de Caralt TM, Ortiz JT, Fita G, Sitges M, Brugada J, Mont L, Berruezo A. Infarct transmurality as a criterion for first-line endo-epicardial substrate-guided ventricular tachycardia ablation in ischemic cardiomyopathy. Heart Rhythm. 2016 Jan;13(1):85-95. doi: 10.1016/j.hrthm.2015.07.010. Epub 2015 Jul 9. PMID 26165946
- [Background] Soto-Iglesias D, Acosta J, Penela D, Fernandez-Armenta J, Cabrera M, Martinez M, Vassanelli F, Alcaine A, Linhart M, Jauregui B, Efimova E, Perea RJ, Prat-Gonzalez S, Ortiz-Perez JT, Bosch X, Mont L, Camara O, Berruezo A. Image-based criteria to identify the presence of epicardial arrhythmogenic substrate in patients with transmural myocardial infarction. Heart Rhythm. 2018 Jun;15(6):814-821. doi: 10.1016/j.hrthm.2018.02.007. Epub 2018 Feb 7. PMID 29427821
- [Background] Fernandez-Armenta J, Penela D, Acosta J, Andreu D, Evertz R, Cabrera M, Korshunov V, Vassanelli F, Martinez M, Guasch E, Arbelo E, Maria Tolosana J, Mont L, Berruezo A. Substrate modification or ventricular tachycardia induction, mapping, and ablation as the first step? A randomized study. Heart Rhythm. 2016 Aug;13(8):1589-95. doi: 10.1016/j.hrthm.2016.05.013. Epub 2016 May 12. PMID 27180621
- [Background] Acosta J, Andreu D, Penela D, Cabrera M, Carlosena A, Korshunov V, Vassanelli F, Borras R, Martinez M, Fernandez-Armenta J, Linhart M, Tolosana JM, Mont L, Berruezo A. Elucidation of hidden slow conduction by double ventricular extrastimuli: a method for further arrhythmic substrate identification in ventricular tachycardia ablation procedures. Europace. 2018 Feb 1;20(2):337-346. doi: 10.1093/europace/euw325. PMID 28017938
- [Background] Berruezo A, Fernandez-Armenta J, Andreu D, Penela D, Herczku C, Evertz R, Cipolletta L, Acosta J, Borras R, Arbelo E, Tolosana JM, Brugada J, Mont L. Scar dechanneling: new method for scar-related left ventricular tachycardia substrate ablation. Circ Arrhythm Electrophysiol. 2015 Apr;8(2):326-36. doi: 10.1161/CIRCEP.114.002386. Epub 2015 Jan 12. PMID 25583983
- [Derived] Falasconi G, Penela D, Soto-Iglesias D, Francia P, Teres C, Viveros D, Bellido A, Alderete J, Meca-Santamaria J, Franco P, Ordonez A, Diaz-Escofet M, Matiello M, Maldonado G, Scherer C, Huguet M, Camara O, Ortiz-Perez JT, Marti-Almor J, Berruezo A. Preventive substrate ablation in chronic post-myocardial infarction patients with high-risk scar characteristics for ventricular arrhythmias: rationale and design of PREVENT-VT study. J Interv Card Electrophysiol. 2023 Jan;66(1):39-47. doi: 10.1007/s10840-022-01392-w. Epub 2022 Oct 13. PMID 36227461